CLINICAL TRIAL: NCT02520869
Title: Diagnostic Value of Sperm DNA Fragmentation and Sperm Morphology for Predicting Outcome of Assisted Reproduction Treatment
Brief Title: Diagnostic Value of Sperm DNA Fragmentation and Sperm Morphology for Assisted Reproduction Treatment
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: khalid abd aziz mohamed (Other)
Responsible Party: Sponsor-Investigator, khalid abd aziz mohamed, lecutrer, Benha University
Organization: Benha University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: wagdy 1
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Assisted Reproductive Technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- swim-up (Active Comparator): swim-up technique for semen processing
  Interventions: Procedure: swim-up technique
- zeta test (Active Comparator): zeta test technique for semen processing
  Interventions: Procedure: zeta test technique

INTERVENTIONS:
Procedure: swim-up technique — swim-up technique used
  Arms: swim-up
Procedure: zeta test technique — zeta test technique used
  Arms: zeta test

SUMMARY:
All patients will go through an ICSI (intracytoplasmic sperm injection)cycle Monitoring: COH (controlled ovarian hyperstimulation) will be monitored by transvaginal sonography, and then the dose of gonadotropin will be adjusted according to the follicle size and number.

Triggering ovulation: when three or more follicles reach >18mm, endometrium triple line >8mm, both the gonadotropin and agonist injections will be stopped and 10,000 IU of hCG(human chorionic gonadotropin ) will be given.

Egg collection : 34-36 hour after hCG injection, embryo transfer :48-72 hour after oocyte retrieval. Luteal phase support: with 100 mg progesterone injection IM daily until the day of the pregnancy test pregnancy test: 15 days after the embryo transfer. Semen collection and preparation Semen samples will be collected by masturbation in clean containers, usually after 2-3 days of abstinence. Each sample will be allowed to liquefy for at least 20 min at 37 °C.

Semen analysis:

Basic sperm parameters including sperm count, concentration, motility and morphology will be evaluated according to World Health Organization guidelines. After the initial assessment, ejaculates will be divided into three aliquots. An aliquot of each sample will be used to assess sperm DNA damage, the second aliquot will be processed by direct swim-up technique (n 30) or zeta test technique (n 30) this will be followed by assessment of DNA damage again in each sample to measure the difference in DNA damage after processing in each technique then spermatozoa from the third aliquot will be morphologically analyzed manually using Spermic stain and a light microscope and will be scored according to WHO

DETAILED DESCRIPTION:
This study will be carried out in private centers for IVF. The aim of this study is to determine the prognostic value of sperm DNA fragmentation levels before and after semen processing and sperm morphology in predicting the outcome of assisted reproduction.

60 couples will undergo ICSI cycles in private centers for IVF. All patients will go through an ICSI cycle. Monitoring: COH will be monitored by transvaginal sonography, and then the dose of gonadotropin will be adjusted according to the follicle size and number.

Triggering ovulation: when three or more follicles reach >18mm, endometrium triple line more than 8mm, both the gonadotropin and agonist injections will be stopped and 10,000 IU of hCG will be given.

Egg collection : 34-36 hour after hCG injection, embryo transfer :48-72 hour after oocyte retrieval. Luteal phase support: with 100 mg progesterone injection intramuscularly daily until the day of the pregnancy test.

pregnancy test: 15 days after the embryo transfer. Semen collection and preparation. Semen samples will be collected by masturbation in clean containers, usually after 2-3 days of abstinence. Each sample will be allowed to liquefy for at least 20 min at 37 °C.

Semen analysis:

Basic sperm parameters including sperm count, concentration, motility and morphology will be evaluated according to World Health Organization guidelines . After the initial assessment, ejaculates will be divided into three aliquots. An aliquot of each sample will be used to assess sperm DNA damage, the second aliquot will be processed by direct swim-up technique (n 30) or zeta test technique (n 30) this will be followed by assessment of DNA damage again in each sample to measure the difference in DNA damage after processing in each technique then spermatozoa from the third aliquot will be morphologically analyzed manually using Spermic stain and a light microscope and will be scored according to WHO.

DNA fragmentation assay:

The assessment of DNA damage will be measured before and after processing for each sample using an improved version of the sperm chromatin dispersion test. Samples will be prepared for analysis. staining step will be required to evaluate the prepared slides. The samples will be stained with Diff-Quik solution, immersing each slide in Diff-Quik solution I (eosinophilic) and Diff-Quik solution II (basophilic) for 6 min each, allowed to dry at room temperature .then the slide will be examined under bright field microscope.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent for the ICSI treatment
* Female body mass index of 18-30 kg/m2
* No congenital uterine anomalies in gynecological ultrasound of female partner
* Male partner not under pharmacological treatment
* couples undergoes ICSI procedures with ejaculated sperm will be included and - Sperm count not less than 0.1 Million per ML
* Male abstinence period 2-3 days.

Exclusion Criteria:

* women over 42 years old
* acute infectious diseases
* systemic illnesses
* Treatment cycles that will result in a poor ovarian response (<3 mature oocytes collected) or those involving epididymal, testicular and cryopreserved sperm samples
* Male patients having varicocele, oligospermia
* male partner under pharmacological treatment

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of spermatozoa with fragmented DNA before and after processing | after taking semen sample by 30 minutes
  Semen samples will be collected by masturbation in clean containers, usually after 2-3 days of abstinence

SECONDARY OUTCOMES:
reproductive success | pregnancy test done 15 days after the embryo transfer.
  by measuring HCG in the patient seruum

CONTACTS AND LOCATIONS:
Overall Officials: wagdy amer, MD, Principal Investigator — lecturer; abo baker el nashar, MD, Study Chair — professor
Locations (1):
- Benha Faculty of Medicine, Banhā, El Qaluobia, Egypt